CLINICAL TRIAL: NCT02106559
Title: A Pilot Study of Pleural Photodynamic Therapy for Patients With Pleural Malignancy
Brief Title: Photodynamic Therapy During Surgery in Treating Patients With Pleural Malignancy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Meng Welliver, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-12223; NCI-2014-00637 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-04-01; First posted 2014-04-08 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Stage III Malignant Mesothelioma; Stage IIIB Non-small Cell Lung Cancer; Stage IV Malignant Mesothelioma; Stage IV Non-small Cell Lung Cancer
Keywords: Pleural Photodynamic Therapy; Pleural Malignancy; PDT
MeSH Terms: conditions — Mesothelioma, Malignant; Carcinoma, Non-Small-Cell Lung | interventions — Dihematoporphyrin Ether; Trioxsalen; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (surgery, porfimer sodium, PDT) (Experimental): Patients receive porfimer sodium IV over 3-5 minutes. Beginning 24 hours later, patients undergo tumor resection and/or radical pleurectomy followed by intraoperative photodynamic therapy to the pleural space.
  Interventions: Drug: porfimer sodium; Procedure: therapeutic conventional surgery; Drug: photodynamic therapy

INTERVENTIONS:
Drug: porfimer sodium — Given IV
  Other Names: CL-184116; DHE; dihematoporphyrin ether; Photofrin II
Procedure: therapeutic conventional surgery — Undergo tumor resection and/or radical pleurectomy
Drug: photodynamic therapy — Undergo PDT
  Other Names: Light Infusion Therapy™; PDT; therapy, photodynamic

SUMMARY:
This pilot clinical trial studies photodynamic therapy during surgery in treating patients with pleural (the protective lining or membrane that covers the lungs and chest cavity) malignancy. Photodynamic therapy is an anti-cancer treatment that combines a photosensitizer (a substance that makes cells more sensitive to light), such as porfimer sodium, together with oxygen and visible light to kill tumor cells and/or damage the tumor's blood supply. Intraoperative (during surgery) photodynamic therapy may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES; I. To determine the feasibility and toxicities of incorporating surgical resection and intra-operative Photofrin (porfimer sodium)-mediated photodynamic therapy in patients (pts) with malignant pleural mesothelioma (MPM) or non-small cell lung cancer (NSCLC) with pleural spread.

SECONDARY OBJECTIVES:

I. To determine the overall survival rate of pts with NSCLC and pleural spread treated with standard frontline chemotherapy followed by surgical resection and intra-operative Photofrin-mediated photodynamic therapy.

II. To determine the overall survival rate of pts with MPM after radical pleurectomy and intraoperative Photofrin-mediated photodynamic therapy (PDT).

III. To determine the progression-free survival and pleural progression-free survival in the above mentioned pts.

IV. To determine the absolute Photofrin levels in tumor and normal tissues resected from pts using spectrofluorometric assay. Photofrin levels in tumor to normal tissue ratios will be determined.

OUTLINE:

Patients receive porfimer sodium intravenously (IV) over 3-5 minutes. Beginning 24 hours later, patients undergo tumor resection and/or radical pleurectomy followed by intraoperative PDT to the pleural space.

After completion of treatment, patients are followed up at 3, 6, 9, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of NSCLC or MPM; pts must have clinical and/or pathological evidence of pleural spread or stage III/IV MPM
* Pts with NSCLC who have received, are receiving or are planning to receive two to four cycles of standard frontline chemotherapy are eligible; choice of chemotherapy is at the discretion of the medical oncologist; concurrent chemoradiotherapy will not be permitted during the active study period; post-operative radiotherapy can be administered as clinically indicated
* Assessment by the attending thoracic surgeon that the primary tumor is resectable in pts with NSCLC and pleural spread; tumor will be deemed resectable if there is no extension through fascia, no bony chest or vertebral body involvement, and no radiographic evidence of mediastinal involvement
* Assessment by the attending thoracic surgeon that radical pleurectomy can be safely achieved in pts with malignant pleural mesothelioma
* All studies required for evaluation will be performed within 8 weeks of Photofrin administration
* Pts of all ethnic and gender groups will be included; protocol accrual will be reviewed annually to include a determination of minority and gender representation; if accrual demonstrates under-representation of any group with comparison to disease incidence in that group, then appropriate measures will be undertaken to attempt to increase participation of pts of that minority or gender group
* ELIGIBILITY CRITERIA FOR HISTORICAL CONTROL POPULATION
* Pts undergoing extrapleural pneumonectomy without PDT for MPM or stage IV (M1A) NSCLC (after American Joint Committee on Cancer [AJCC] staging change 2010) or stage IIIB (before staging change) with malignant pleural effusion treated at Ohio State University (OSU) from 2005-2012
* Historical control data will be derived from patient medical records at the Ohio State University Medical Center (OSUMC)

Exclusion Criteria:

* Pts who have grade III-IV elevations in liver transaminases (as defined by the Common Terminology Criteria for Adverse Events [CTCAE] version [v.] 4.0) or a bilirubin in excess of 1.5 mg/dl
* Pts who are medically unfit to tolerate surgery
* Pts with known human immunodeficiency virus (HIV) or hepatitis C virus (HCV) disease (routine testing is not needed if not clinical indicated)
* Pregnant or lactating pts
* Prior treatment for NSCLC except for pleurodesis and/or standard frontline chemotherapy
* Pts who have received prior mantle or extensive mediastinal radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2016-01-29 (Actual); Study Completion 2016-01-29 (Actual)

PRIMARY OUTCOMES:
Number of patients who received the entire multi-modality regimen | Up to 2 years
Incidence of grade 4 or greater toxicity in the post-operative period as graded by the National Cancer Institute (NCI) CTCAE (Common Toxicity Criteria for Adverse Effects) version 4.0 | Up to 90 days post surgery
  All observed toxicities will be graded, tabled and summarized by frequencies and percentages.

SECONDARY OUTCOMES:
Overall survival | Time from study entry (start of chemotherapy) to death due to any cause or last patient contact, assessed up to 2 years
  Estimated by the method of Kaplan and Meier. Overall survival will be estimated for all patients entered on trial, regardless of treatment received on-study or off-study.
Progression-free survival (PFS) | Time from study entry to first documented progression (any type, intrapleural, distant, locoregional) or death due to any cause, assessed up to 2 years
  Estimated by the method of Kaplan and Meier. PFS will be estimated for all patients entered on trial, regardless of treatment received on-study or off-study.
Pleural progression-free survival (PPFS) | Time from surgery/PDT to first documented intrapleural progression or death from any cause, assessed up to 2 years
  Estimated by the method of Kaplan and Meier. PPFS will be estimated for the subset of patients who receive PDT, in order to evaluate the impact of PDT on local control. Survival curves will be plotted. Median and 1-year estimates and confidence intervals will be calculated.
Porfimer sodium uptake defined as the ratio of the porfimer sodium concentration in tumor tissue to normal tissue (i.e. skin) using spectrofluorometric assay | After surgery
  Porfimer sodium concentration in the tissue will be calculated based on the increase in fluorescence resulting from the addition of a known amount of porfimer sodium to each sample after its initial reading. Absolute concentrations of porfimer sodium will also be measured. Distribution of uptake will be summarized by mean, median, standard deviation, range, and histogram. The tumor: normal tissue ratio from direct and indirect measurements will be calculated. Spearman's correlation will be employed to correlate and compare direct and indirect measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Welliver, Principal Investigator — Ohio State University Comprehensive Cancer Center

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu